CLINICAL TRIAL: NCT04776005
Title: Multicenter, Observational Study of Anti-Sars-Cov2 Vaccine Efficacy in Patients With Malignant Pathologies Treated in the University Hospitals of AP-HP. Nord
Brief Title: COVID-19 Vaccine Efficacy in Patients With Malignant Pathologies
Acronym: COVIDVAC OH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210640
Record Dates: First submitted 2021-02-26; First posted 2021-03-01 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Solid Tumor; Hematologic Malignancy; Thoracic Cancer; Cancer, Treatment-Related; Vaccine Response Impaired
Keywords: Malignant pathology; Hematologic malignancy; COVID-19; Vaccine; Sars-CoV-2 antibody
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms, Second Primary; COVID-19 | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Patients with malignant disease undergoing chemotherapy: Patients with malignant disease undergoing chemotherapy within the University Hospital Centre AP-HP.Nord, who have voluntarily agreed to be vaccinated with an approved vaccine against the Sars-CoV-2 virus.
  Interventions: Other: Data collection
- Patients with malignant disease undergoing chemotherapy + immunotherapy: Patients with malignant disease undergoing chemotherapy + immunotherapy within the University Hospital Centre AP-HP.Nord, who have voluntarily agreed to be vaccinated with an approved vaccine against the Sars-CoV-2 virus.
  Interventions: Other: Data collection
- Patients with malignant disease undergoing immunotherapy: Patients with malignant disease undergoing immunotherapy within the University Hospital Centre AP-HP.Nord, who have voluntarily agreed to be vaccinated with an approved vaccine against the Sars-CoV-2 virus.
  Interventions: Other: Data collection
- Patients with malignant disease treated with targeted therapies: Patients with malignant disease treated with targeted therapies within the University Hospital Centre AP-HP.Nord, who have voluntarily agreed to be vaccinated with an approved vaccine against the Sars-CoV-2 virus.
  Interventions: Other: Data collection
- Patients with malignant disease undergoing radiotherapy: Patients with malignant disease undergoing radiotherapy within the University Hospital Centre AP-HP.Nord, who have voluntarily agreed to be vaccinated with an approved vaccine against the Sars-CoV-2 virus.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Assessment of the efficacy and immunogenicity of the anti-Sars-COv2 vaccines in patients treated for malignant pathology.

SUMMARY:
In the context of malignant disease, it is likely that vaccine efficacy and immunogenicity depends on the type of pathology, stage of the disease, immunosuppression induced by the treatments, in addition to more classic factors such as age, general condition and possibly the type of vaccine used.

There are very little data on the efficacy and immunogenicity of anti-severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines in patients with malignant disease in the active phase of treatment.

This multicenter observational study aims to assess the efficacy and the immunogenicity of anti-Sars-CoV-2 vaccines in the cohort of patients treated for malignant pathology (solid or hematological tumors) at Saint Louis Hospital and in thoracic oncology patients at Bichat Hospital.

DETAILED DESCRIPTION:
During the visit carried out as part of the follow-up, participation in this study will be proposed to any patient who is treated for a malignant disease (solid or hematological tumors) within the university hospitals of AP-HP.Nord.

The patients participating in this prospective cohort will benefit from all standard care his/her condition requires.

Clinical and biological data will be collected as part of the usual follow-up. Clinical data: pathology, stage, treatment line, type of current treatment and date of the last treatment administered, previous treatments, radiotherapy, concept of radiation lung disease, history of pneumonectomy, comorbidities, performance status, history of coronavirus disease 2019 (COVID-19).

Laboratory data: pre-vaccination polynuclear neutrophil count, lymphocyte counts, plasma protein electrophoresis or Ig weight dosage (routine care in hematology), lactate dehydrogenase (LDH), C-reactive protein (CRP), albuminemia in the previous month.

Vaccination data: type of vaccine, date of the 1st injection, date of the 2nd injection, pre-vaccination antibody levels

* Seroconversion with anti-S IgG after anti-Sars-CoV-2 vaccination
* Anti-S and / or anti-N Sars-CoV-2 IgG seroprevalence before vaccination
* Adverse effects related to vaccines
* Levels of the anti-S IgG antibodies in AU / ml

During visits between D21 and D28 (before the 2nd injection), at month 3, month 6 and month 12, the following data will be collected:

* Antibody levels
* Adverse effects related to vaccines
* Levels of the anti-S IgG antibodies in AU / ml
* Associated side effects
* Occurrence of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant disease undergoing treatment at Saint Louis Hospital or Bichat Hospital (for chest cancer)
* with chemotherapy
* with chemotherapy + Immunotherapy
* with immunotherapy
* with targeted therapies
* with radiotherapy
* in the event of radiation pneumonitis after radiotherapy for lung cancers
* after pneumonectomy for lung cancer
* Patient informed and having expressed their non-opposition to participating in this research

Exclusion Criteria:

* Patient with a contraindication to Sars-Cov2 vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are treated for a malignant disease (solid or hematological tumors) within the CHU AP-HP.Nord and who are willing to get a SARS-CoV-2 vaccination.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 vaccine response at 12 months | 12 months
  IgG anti-Sarc-CoV-2 S-protein titer at 12 months

SECONDARY OUTCOMES:
Seroprevalence of antibodies against Sarc-CoV-2 S-protein before vaccination | Day 0
  Rate of patients presenting the anti Sarc-CoV-2 S-protein antibodies before vaccination in the study population.
Seroprevalence of antibodies against Sarc-CoV-2 N-protein before vaccination | Day 0
  Rate of patients presenting the anti Sarc-CoV-2 N-protein antibodies before vaccination in the study population.
SARS-CoV-2 vaccine response after first dose of vaccine | Day 24 +/- 4 days
  IgG anti-Sarc-CoV-2 S-protein titer after the first injection of vaccine
SARS-CoV-2 vaccine response at 3 months | 3 months
  IgG anti-Sarc-CoV-2 S-protein titer at 3 months
SARS-CoV-2 vaccine response at 6 months | 6 months
  IgG anti-Sarc-CoV-2 S-protein titer at 6 months
SARS-CoV-2 vaccine safety in the study population | 12 months
  Occurence of the adverse events related to the SARS-CoV-2 vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Luis TEIXEIRA, MD, PhD, Principal Investigator — Breast Disease Unit, Saint-Louis Hospital, APHP, Université de Paris, INSERM U976
Locations (2):
- France (2):
  - Saint-Louis Hospital, AP-HP, Paris
  - Bichat Hospital, AP-HP, Paris

IPD SHARING:
Plan to Share IPD: Undecided